CLINICAL TRIAL: NCT02670044
Title: A Phase IB Multi-Arm Study With Venetoclax in Combination With Cobimetinib and Venetoclax in Combination With Idasanutlin in Patients With Relapsed or Refractory Acute Myeloid Leukemia Who Are Not Eligible for Cytotoxic Therapy
Brief Title: A Study of Venetoclax in Combination With Cobimetinib and Venetoclax in Combination With Idasanutlin in Patients With Relapsed or Refractory Acute Myeloid Leukemia Who Are Not Eligible for Cytotoxic Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH29914; 2015-003386-28 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cobimetinib; RG7388; venetoclax

ARMS (9):
- Dose Escalation: Arm A (Venetoclax 400mg + Cobi 40mg) (Experimental): Participants received Venetoclax 400mg daily on Days 1-28 of each 28 day treatment cycle and Cobimetinib 40mg daily on Days 1-21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- Dose Escalation: Arm A (Venetoclax 600mg + Cobi 40mg) (Experimental): Participants received Venetoclax 600mg daily on Days 1-28 of each 28 day treatment cycle and Cobimetinib 40mg daily on Days 1-21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- Dose Escalation: Arm A (Venetoclax 800mg + Cobi 40mg) (Experimental): Participants received Venetoclax 800mg daily on Days 1-28 of each 28 day treatment cycle and Cobimetinib 40mg daily on Days 1-21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- Dose Escalation: Arm A (Venetoclax 400mg + Cobi 60mg) (Experimental): Participants received Venetoclax 400mg daily on Days 1-28 of each 28 day treatment cycle and Cobimetinib 60mg daily on Days 1-21 of each 28-day treatment cycle.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- Dose Escalation: Arm B (Venetoclax 400mg + Ida 200mg) (Experimental): Participants received Venetoclax 400mg daily on Days 1-28 of each 28 day treatment cycle and Idasanutlin 200mg daily or twice daily on Days 1-5 of each 28 day treatment cycle.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax
- Dose Escalation: Arm B (Venetoclax 600mg + Ida 150mg) (Experimental): Participants received Venetoclax 600mg daily on Days 1-28 of each 28 day treatment cycle and Idasanutlin 150mg daily or twice daily on Days 1-5 of each 28 day treatment cycle.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax
- Dose Escalation: Arm B (Venetoclax 600mg + Ida 200mg) (Experimental): Participants received Venetoclax 600mg daily on Days 1-28 of each 28 day treatment cycle and Idasanutlin 200mg daily or twice daily on Days 1-5 of each 28 day treatment cycle.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax
- Dose Escalation: Arm B (Venetoclax 400mg + Ida 400mg) (Experimental): Participants received Venetoclax 400mg daily on Days 1-28 of each 28 day treatment cycle and Idasanutlin 400mg daily or twice daily on Days 1-5 of each 28 day treatment cycle.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax
- Dose Optimisation: Arm B (Ven 600mg (Day 1 to 21) + Ida 150mg) (Experimental): Participants received Venetoclax 600mg daily on Days 1-21 of each 28 day treatment cycle and Idasanutlin 150mg daily on Days 1-5 of each 28 day treatment cycle.
  Interventions: Drug: Idasanutlin; Drug: Venetoclax

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be administered orally as per schedule in Arm description.
  Arms: Dose Escalation: Arm A (Venetoclax 400mg + Cobi 40mg); Dose Escalation: Arm A (Venetoclax 400mg + Cobi 60mg); Dose Escalation: Arm A (Venetoclax 600mg + Cobi 40mg); Dose Escalation: Arm A (Venetoclax 800mg + Cobi 40mg)
Drug: Idasanutlin — Idasanutlin will be administered orally as per schedule in Arm description.
  Arms: Dose Escalation: Arm B (Venetoclax 400mg + Ida 200mg); Dose Escalation: Arm B (Venetoclax 400mg + Ida 400mg); Dose Escalation: Arm B (Venetoclax 600mg + Ida 150mg); Dose Escalation: Arm B (Venetoclax 600mg + Ida 200mg); Dose Optimisation: Arm B (Ven 600mg (Day 1 to 21) + Ida 150mg)
Drug: Venetoclax — Venetoclax will be administered orally as per schedule in Arm description.

SUMMARY:
The primary objective for this study is to assess the safety and tolerability as well as preliminary efficacy of venetoclax in combination with cobimetinib, and venetoclax in combination with idasanutlin in patients with relapsed or refractory acute myeloid leukemia (R/R) AML who are not eligible for cytotoxic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of relapsed or refractory AML after prior anti-leukemic therapy by WHO classification
* Ineligible for cytotoxic therapy defined by the following:

  a. Age (>/=) 75 years or b. age 18- 74 years with at least one of the following comorbidities: i. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3 ii. Cardiac history of congestive heart failure requiring treatment or ejection fraction (</=) 50% or chronic stable angina iii. Diffusing capacity of the lungs for carbon monoxide (</=) 65% or forced expiratory volume in the first second of expiration (</=) 65% iv. Creatinine clearance (>/=) 30 mL/min to< 45 mL/min v. any other comorbidity that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the Medical Monitor before screening and study enrollment.
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Adequate liver and renal function

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (French-American-British [FAB] class M3 AML)
* Known active central nervous system (CNS) involvement with AML at study entry
* ECOG Performance Status (>/=) 3 in patients who are (>/=) 75 years old or ECOG Performance Status of 4, regardless of age
* Prior exposure to Bcl-2 inhibitors, murine double minute 2 (MDM2) antagonists or prior exposure to experimental treatment targeting Raf, mitogen-activated protein kinase (MEK), or the mitogen-activated protein kinase (MAPK) RAS/RAF/MEK/ERK MAPK pathway
* Positive for hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg) and known history of HIV, malignancy, active infection and cardiovascular diseases (CVs)
* Received strong cytochrome (CYP) 3A inhibitors, moderate CYP3A inhibitors, strong CYP3A inducers and moderate CYP3A inducers within 7 days prior to initiation of study treatment
* History of symptomatic Clostridium difficile infection within 1 month prior to dosing

Additional arm specific exclusion criteria:

Dose Escalation Arm A (Venetoclax and Cobimetinib):

* History or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower

Arm B (Venetoclax and Idasanutlin):

* Received the following within 7 days prior to the initiation of study treatment: Strong CYP2C8 inhibitors or CYP2C8 substrates, OATP1B1/3 substrates
* Received the following within 14 days prior to the initiation of study treatment: Strong CYP2C8 inducers
* History of liver cirrhosis by radiologic, clinical or laboratory data, or biopsy despite normal liver function tests
* Received treatment with oral or parenteral anticoagulants/anti-platelet agents within 7 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | From Cycle 1 Day 1 to Cycle 2 Day 1 for a minimum of 28 days
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Baseline up until 30 days after the last dose of study drug (up to a maximum of 4 years, 9 months)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) (Complete Remission (CR) + Complete Remission with Incomplete Blood Recovery (CRi) + Incomplete Platelet Count Recovery (CRp) + Partial Remission/Partial Response [PR]) | Up to 2 years
Complete Remission/complete response (CR) + Complete Remission with Incomplete Blood Recovery (CRi) + Incomplete Platelet Count Recovery (CRp) | Up to 2 years
CR + Complete Remission with Partial Hematologic Recovery (CRh) Rate | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Time to Progression (TTP) | Up to 2 years
Progression-Free Survival (PFS) | Up to 2 years
Event-Free Survival (EFS) | Up to 2 years
Leukemia-Free Survival (LFS) | Up to 2 years
Overall Survival (OS) | Up to 2 years
Pharmacokinetics of Venetoclax Area Under the Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-24hr) | Up to 6 months
Pharmacokinetics of Venetoclax Maximum Observed Concentration (Cmax) | Up to 6 months
Pharmacokinetics of Cobimetinib Area Under the Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-24hr) | Up to 6 months
Pharmacokinetics of Cobimetinib Maximum Observed Concentration (Cmax) | Up to 6 months
Pharmacokinetics of Idasanutlin Area Under the Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-24hr) | Up to 6 months
Pharmacokinetics of Idasanutlin Maximum Observed Concentration (Cmax) | Up to 6 months
Number of Participants Reporting Symptoms in Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Questionnaire | Up to 2 years
Rate of Transfusion Independence | Up to 2 years
Duration Of Transfusion Independence, Defined As The Number Of Consecutive Days Of Transfusion Independence, Measured From 1 Day After Last Transfusion To Disease Progression Or Subsequent Transfusion | Up to 2 years
Minimal Residual Disease (MRD) In The Bone Marrow To Evaluate The Depth Of Response | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (8):
  - USC Norris Cancer Center, Los Angeles, California
  - UC Davis; Comprehensive Cancer Center, Sacramento, California
  - Univ of Calif, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (3):
  - Hopital Avicenne, Paris, Bobigny
  - Institut Paoli Calmettes, Marseille
  - CHU de Bordeaux, Pessac
- Italy (3):
  - University of Bologna, Bologna, Emilia-Romagna
  - Presidio san salvatore muraglia, Pesaro, Emilia-Romagna
  - Universita di Roma, Roma, Emilia-Romagna

REFERENCES:
- [Derived] Daver NG, Dail M, Garcia JS, Jonas BA, Yee KWL, Kelly KR, Vey N, Assouline S, Roboz GJ, Paolini S, Pollyea DA, Tafuri A, Brandwein JM, Pigneux A, Powell BL, Fenaux P, Olin RL, Visani G, Martinelli G, Onishi M, Wang J, Huang W, Green C, Ott MG, Hong WJ, Konopleva MY, Andreeff M. Venetoclax and idasanutlin in relapsed/refractory AML: a nonrandomized, open-label phase 1b trial. Blood. 2023 Mar 16;141(11):1265-1276. doi: 10.1182/blood.2022016362. PMID 36265087